CLINICAL TRIAL: NCT02329509
Title: Evaluation of Facial Growth in Two Primary Protocols Used in the Surgical Treatment of Unilateral Cleft Lip and Palate Patients. A Prospective Randomized Trial
Brief Title: Evaluation of Facial Growth in Two Primary Protocols Used in the Surgical Treatment of Unilateral Cleft Lip and Palate Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rui Manuel Rodrigues Pereira, CADEFI Coordinator, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1158-3755; CADEFI /IMIP (Other: CADEFI/IMIP)
Record Dates: First submitted 2014-12-16; First posted 2014-12-31 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Unilateral Cleft Lip and Palate; Cleft Lip; Cleft Palate; Developmental Disabilities; Restricted Language Development
Keywords: operative procedures
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Developmental Disabilities

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- one stage cleft palate surgery (Active Comparator): Subjects submitted to one stage palate surgical repair after 9 months old and before 24 months old ,
  Interventions: Procedure: One stage Palate Surgical repair
- two stage palate repair (Active Comparator): Subjects submitted to two stage palate surgical repair (first soft palate repair between 6 and 12 months old and hard palate closure at 3 to 4 years old)
  Interventions: Procedure: two stage palate surgical repair

INTERVENTIONS:
Procedure: two stage palate surgical repair — two stage palate surgical repair with a hard palate closure at 3 to 4 years old
  Arms: two stage palate repair
Procedure: One stage Palate Surgical repair — One stage palate repair at the age of 9 to 24 months old
  Arms: one stage cleft palate surgery

SUMMARY:
The purpose of this study is to evaluate which surgical protocol for treating Unilateral Cleft Lip and Palate (UCLP), a single or two stage repair ( with hard palate late closure) will have less impact in mid facial growth.

The study hypothesis states that a two stage cleft palate repair , with a late hard palate repair will reduce maxillary growth impairment.

DETAILED DESCRIPTION:
The study is being conducted at CADEFI- Centro de Atenção aos Defeitos da Face do IMIP (craniofacial center) in IMIP-Instituto de Medicina Integral Professor Fernando Figueira-, Recife PE- Pernambuco-, Brazil. All children were and will be operated by the same plastic surgeon in the operating room in IMIP. The sample size was calculated in 64 patients, 32 to GI ( one stage repair) and 32 to GII ( two stage repair, with a hard palate late closure), considering taking a statistical power of 90% with a 5% significance, determined with a difference of at least 25% between the two groups. Note : this sample was calculated for the dependent variable commonly present in patients with unilateral lip and palate cleft : atresia of the dental arches.

The groups are numbered in post op care attendance of the lip repair, according to randomization sequence done in computerized statistical program. The randomization is being held after the first month of the lip repair surgery. The surgeon, and parents or guardians (who have already signed the Informed Consent Form) will not have prior access to information on the type of allocation in each group. Subsequently it will be added in patients chart the record set for the patient group.

>Study Variables Independent variables:. Group I (palate closure in two surgical times and GII (closure of the palate in a surgical time) also will be considered independent variables age, sex, birth weight and maternal education.

Dependent variables: the presence of postoperative infection, initial and intermediate cleft sizes, dimensional changes of the transverse arch, the evaluation indexes of dental arch relationship(Goslom,Atack Yardsticks) and speech outcomes evaluation grades

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral cleft lip and palate admitted consecutively in CADEFI-IMIP between August 1, 2011 and July 31, 2015

Exclusion Criteria:

* Patients with associated syndromes that retard the neuro-psycho-motor and speech development;
* Patients without clinical conditions for performing the surgical chronology protocol;
* Patients whose parents or guardians who are not in accordance with the Informed Consent Statement proposed by the researcher

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Maxillary Growth Evaluated by the Atack Yardstick | between 4 to 5 years old
  A system that evaluates facial growth , assessing dental arch relationships, and ranking them from 1 to 5, being 1 the best and 5 the worst outcome.Cases are allocated to these categories on a value judgment basis by reference to the anchor groups of the Atack Yardstick. This is performed by external judges, previously trained and evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nivaldo Alonso, PH.D, Study Director — USP